CLINICAL TRIAL: NCT01561794
Title: A Prospective, Non-randomized, Open-label, Non-controlled, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics/ Pharmacodynamics of BAYQ3939 (400 mg BID and TID) in Hospitalized Patients With Bacterial Pneumonia or Secondary Infection of Chronic Respiratory Disease With Severe Disease or a Poor Response to Other Antimicrobials
Brief Title: A Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics/Pharmacodynamics of BAYQ3939 in Patients With Bacterial Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15992
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Pneumonia
Keywords: Ciprofloxacin; Bacterial pneumonia; Community Acquired Pneumonia (CAP); Hospital Acquired Pneumonia (HAP); Secondary infection of chronic respiratory disease; 400 mg BID/TID
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ciprofloxacin (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro, BAYQ3939)

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro, BAYQ3939) — (1) Community-acquired pneumonia (CAP): 400 mg BID, i.e. every 12 ± 1 hours (For those with Ccr > 60 mL/min, 400 mg TID, i.e. every 8 ± 1 hours may be considered at the discretion of investigators) for 7 to 14 days.
  2) Hospital-acquired pneumonia (HAP): For the patient with Ccr > 60 mL/min, 400 mg TID, i.e. every 8 ± 1hours for 7 to 14 days For the patient with 30 ≤Ccr ≤60 mL/min, 400 mg BID, i.e. every 12 ± 1hours for 7 to 14 days 3) Secondary infection of chronic respiratory disease 400 mg BID, i.e. every 12 ± 1 hours (For those with of Ccr > 60 mL/min, 400 mg TID, i.e. every 8 ± 1 hours may be considered at the discretion of investigators) for 7 to 14 days.

SUMMARY:
The main objective of this study is to investigate the safety, pharmacokinetics (PK) and the relationship between PK and pharmacodynamics (Minimum Inhibitory Concentration [MIC] and Mutant Prevention Concentration [MPC]) of intravenous BAYQ3939 (400 mg BID and 400 mg TID) in hospitalized patients with bacterial pneumonia or secondary infection of chronic respiratory disease with severe disease or a poor response to other antimicrobials. In addition, the efficacy of the ciprofloxacin, in terms of clinical response and microbiological response, will be investigated, but as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females with written informed consent, 20 years of age or older.
* Within 48 hours prior to the first study drug administration, all patients should have the pathogens identified with appropriate specimens (e.g., sputum, tracheal aspirate, bronchoalveolar lavage [BAL], protected brushing specimen [PBS]), or should have appropriate specimens highly likely to identify the pathogens sampled. (However, the patients with Legionellosis is enrolled when the test of Legionella antigen is positive.)
* The following severe bacterial pneumonia meeting the diagnostic criteria of pneumonia or secondary infection of chronic respiratory disease

  * Severe pneumonia

    * Community-acquired pneumonia: PORT score III, IV or V
    * Hospital-acquired pneumonia [HAP]-Group B and with a low risk for multidrug-resistant pathogens
    * Patients with [HAP]-Group A whose pathogen is suspected to be Pseudomonas aeruginosa
    * Hospitalized patients with bacterial pneumonia with a poor response to other antimicrobials Note: The patients should be limited to CAP patients with PORT score III, IV or V and HAP patients with-Group A or B who don't respond to or have a poor response to other antimicrobials over 3day's treatment.2
  * Secondary infection of chronic respiratory disease

    * Patients who are hospitalized for the treatment of secondary infection of chronic respiratory disease
    * Hospitalized patients with secondary infection of chronic respiratory disease with a poor response to other antimicrobials Note: The patients should be limited to secondary infection of chronic respiratory disease patients who don't respond to or have a poor response to other antimicrobials over 3day's treatment.

Exclusion Criteria:

* Creatinine clearance (Ccr) ≤ 30 mL/min or nephrotic syndrome
* Patient with chronic treatment of immunosuppressive drug
* Decompensated congestive heart failure
* Subject who received more than 24 hours of an antibacterial drug for the current infection
* Patient who requires Intensive Care Unit (ICU) management [In case subjects who don't correspond to the severity for ICU management need to be admitted to ICU due to a circumstance of the site (e.g. shortage of hospital beds), those subjects shall not be excluded]
* Patients with infections other than pneumonia or secondary infection of chronic pulmonary disease
* Lung abscess, or empyema
* Viral, fungal, mycobacterial, or atypical pneumonia as a primary diagnosis
* Known or suspected bacteremia secondary to Staphylococcus aureus
* Known causative microorganisms other than indication (microorganisms) of the study drug, or positive in urinary antigen test of Streptococcus pneumonia
* Infection that necessitates the use of a concomitant antibacterial agent in addition to study medication [excluding subjects with concomitant use of long-term, low-dose macrolide for chronic respiratory diseases, sulbactam sodium/ampicillin sodium (Unasyn-S) and clindamycin (Dalacin-S)]
* Known bronchial obstruction or a history of post-obstructive pneumonia
* Known primary lung cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | Up to 30 (±5) days after the end of treatment
AUC (Area under the blood concentration/time curve) | Within 0-24 hours and 48-72 hours after the first study drug administration
Cmax (Maximum observed concentration) | Within 0-24 hours and 48-72 hours after the first study drug administration
AUC/MIC (Minimum inhibitory concentration) | Within 0-24 hours and 48-72 hours after the first study drug administration
Cmax/MIC | Within 0-24 hours and 48-72 hours after the first study drug administration
AUC/MPC (Mutant prevention concentration) | Within 0-24 hours and 48-72 hours after the first study drug administration
Cmax/MPC | Within 0-24 hours and 48-72 hours after the first study drug administration

SECONDARY OUTCOMES:
Clinical response rate based on resolution of signs and symptoms | Up to 13 days after the first study drug administration
Microbiological response rate, assessed as eradication rate based on microbiologically evaluable patients | Up to 23 days after the first study drug administration
Test of cure rate based on resolution of signs, symptoms, and the clinical response | Up to 23 days after the first study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Japan (15):
  - Nagakute, Aichi-ken
  - Kobe, Hyōgo
  - Kahoku-gun, Ishikawa-ken
  - Yokohama, Kanagawa
  - Isahaya, Nagasaki
  - Nagasaki, Nagasaki
  - Sasebo, Nagasaki
  - Unzen, Nagasaki
  - Niigata, Niigata
  - Yufu, Oita Prefecture
  - Okayama, Okayama-ken
  - Kishiwada, Osaka
  - Osaka, Osaka
  - Ureshino, Saga-ken
  - Hamamatsu, Shizuoka